CLINICAL TRIAL: NCT02280941
Title: Comparison of Myocardial Blood Flow Measurements With Dedicated Solid State SPECT Camera Imaging and 99mTc-Tetrofosmin Versus PET Imaging and Rubidium-82
Brief Title: Cadmium-zinc-telluride (CZT) Imaging of Myocardial Blood Flow (MBF) (SPECT MBF)
Acronym: SPECTMBF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20140589
Record Dates: First submitted 2014-10-07; First posted 2014-11-03 (Estimated); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-01

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single photon emission computed tomography (Experimental): Myocardial blood flow (MBF) measurement will be analyzed using attenuation and scatter corrected dynamic single photon emission computed tomography (SPECT) imaging data. The data will be compared to MBF obtained from positron emission tomography (PET) imaging.
  Interventions: Other: single photon emission computed tomography

INTERVENTIONS:
Other: single photon emission computed tomography — Single photon emission computed tomography (SPECT) imaging will be done.

SUMMARY:
This study is being done to compare the blood flow measurements obtained with the SPECT and PET imaging scans. Measurements such as myocardial blood flow (MBF) and myocardial flow reserve (MFR) are analyzed on PET scans. These measurements give the doctors more precise information in diagnosing heart problems. SPECT scans, with new camera technology and computer software, now have the potential to also give this additional information. The study is investigating how well the blood flow measurements from SPECT compared to PET.

DETAILED DESCRIPTION:
Absolute myocardial blood flow (MBF) and myocardial flow reserve (MFR) are calculated measurements that are obtained using positron emission tomography (PET) nuclear imaging, from a myocardial perfusion imaging (MPI) stress test, due to the advanced capabilities of the PET camera technology. These calculations provide more diagnostic and prognostic information for patients. Single photon emission computed tomography (SPECT) nuclear imaging is more widely done due to the availability and lower costs, but in the past has not been able to provide the additional information needed to perform the MBF and MFR calculations. SPECT cameras have now been developed and are in use, as well as software for the cameras that have shown that these measurements can be obtained from SPECT. The goal of this study is to compare SPECT and PET measurement of MBF and MFR and determine the reproducibility of SPECT MFR measurements.

The study will be done in 3 Phases, with recruitment done over 3 years. Phase 1 and 2 will be done over the first 2 years, with Phase 3 planned following Phases 1 and 2, in the 3rd year of recruitment.

Phase 1: patients with coronary artery disease, who are coming to the University of Ottawa Heart Institute (UOHI) for MPI stress testing will have both a PET and SPECT MPI for comparison of the measurements of MBF and MFR. The PET scan will be done as the clinical, reportable test.

Phase 2: patients with coronary artery disease, who are coming to UOHI for SPECT MPI testing will have the SPECT repeated to see how reproducible the measurements are.

Phase 3: normal, healthy volunteers will have both a PET and SPECT scan for the comparison of the measurements of MBF and MFR.

No change to any patient care will be done in Phases 1 and 2. Phase 1 and Phase 2 participants will have 1 research scan and Phase 3 participants will have 2 research scans.

Rubidium (Rb-82) Elution System Performance Data will be collected on the elution pump system, used to deliver the Rb-82 isotope, to support the system performance documentation for Health Canada Authorization.

ELIGIBILITY:
Inclusion Criteria:

For all participants

* Age ≥ 18 years old
* BMI ≤ 40 kg/m2
* Able and willing to comply with the study procedures
* Written informed consent Participants with intermediate to high probability of CAD
* Suspected or known CAD on a stable medication regime. Healthy volunteers without known heart disease
* Low risk of CAD (ACC Guidelines Pre-test Probability of Coronary Disease by Symptoms, Gender and Age)

Exclusion Criteria:

* History or risk of severe bradycardia (heart rate < 50 beats per minute) not related to chronotropic drugs
* Known second- or third-degree AV block without pacemaker
* Dyspnea (NYHA III/IV), wheezing asthma or COPD
* Coronary artery bypass graft (CABG) surgery within 60 days prior to screening or at any time after consent
* Percutaneous coronary intervention (PCI) within 30 days prior to screening or at any time following consent
* Acute myocardial infarction or acute coronary syndrome within 60 days prior to screening or at any time following consent
* Recent use of dipyridamole, dipyridamole-containing medications (e.g. Aggrenox)
* Known hypersensitivity to dipyridamole
* Breastfeeding or pregnancy
* Claustrophobia or inability to lie still in a supine position
* Unwillingness or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wells RG, Marvin B, Poirier M, Renaud J, deKemp RA, Ruddy TD. Optimization of SPECT Measurement of Myocardial Blood Flow with Corrections for Attenuation, Motion, and Blood Binding Compared with PET. J Nucl Med. 2017 Dec;58(12):2013-2019. doi: 10.2967/jnumed.117.191049. Epub 2017 Jun 13. PMID 28611245
- [Result] Do J, Ruddy TD, Wells RG. Reduced acquisition times for measurement of myocardial blood flow with 99mTc-tetrofosmin and solid-state detector SPECT. J Nucl Cardiol. 2021 Dec;28(6):2518-2529. doi: 10.1007/s12350-020-02048-w. Epub 2020 Feb 5. PMID 32026329
- [Result] Wells RG, Radonjic I, Clackdoyle D, Do J, Marvin B, Carey C, deKemp RA, Ruddy TD. Test-Retest Precision of Myocardial Blood Flow Measurements With 99mTc-Tetrofosmin and Solid-State Detector Single Photon Emission Computed Tomography. Circ Cardiovasc Imaging. 2020 Feb;13(2):e009769. doi: 10.1161/CIRCIMAGING.119.009769. Epub 2020 Feb 11. PMID 32069116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited 32 patients with known coronary artery disease. Patients were recruited from diagnostic clinic lists.
Pre-assignment Details: Enrolled patients who underwent CABG or PCI after they provided consent were excluded from the study. Enrolled patients who experienced acute myocardial infarction or acute coronary syndrome any time after the consent, were also excluded. Enrolled patients with a positive pregnancy screen prior to their research scan were excluded from the study.
Period: Overall Study
Arm/Group | Single Photon Emission Computed Tomography
Started | 32
Completed | 31
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Photon Emission Computed Tomography
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 31
Suspected or known coronary artery disease [Count of Participants; unit: Participants] | 31

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Measurements of Myocardial Blood Flow Measured With PET and With SPECT
Description: PET studies were acquired with either 82Rb or 13N-ammonia according to clinical protocol. The activity injected at both rest and stress was 10 MBq/kg (82Rb) or 5MBq/kg (ammonia). MBF was based on data acquired over 8 min (82Rb) or 4 min (ammonia). SPECT rest images were obtained for 11 min starting immediately before injection of 316 +/- 71 MBq of 99mTc-tetrofosmin. The patient returned at 45 min after injection for a 5 min static resting acquisition (corresponding to the standard time for myocardial perfusion imaging). Without repositioning, the patient was stressed using dipyridamole (0.14mg/kg/min for 5 minutes) with 11 minutes of list mode data acquired starting immediately before the injection of 1122 +/- 170 MBq of tetrofosmin. Both rest and stress injections were delivered mechanically over 30 seconds. A standard set of stress perfusion images were acquired at 45 mins after tracer injection. The myocardial blood flow obtained using SPECT was compared to the patient's PET.
Time Frame: From enrollment to completion of imaging was a maximum of four weeks. The average difference in acquisition dates was 19 +/- 9 days.
Population: Patients with known coronary artery disease who underwent both PET and SPECT myocardial perfusion imaging within 4 weeks.
Measure: Mean (Standard Deviation); unit: mean residual difference in MBF
Groups:
- Comparision of Myocardial Blood Flow Between PET to SPECT Myocardial Perfusion Imaging.: Myocardial blood flow (MBF) measurement was analyzed using attenuation and scatter corrected dynamic single photon emission computed tomography (SPECT) imaging data. The data will be compared to MBF obtained from positron emission tomography (PET) imaging.
  PET studies were acquired with either 82Rb or 13N-ammonia according to clinical protocol. The activity injected at both rest and stress was 10 MBq/kg (82Rb) or 5MBq/kg (ammonia). MBF was based on data acquired over 8 min (82Rb) or 4 min (ammonia). SPECT rest images were obtained for 11 min starting immediately before injection of 316 +/- 71 MBq of 99mTc-tetrofosmin. The patient returned at 45 min after injection for a 5 min static resting acquisition (corresponding to the standard time for myocardial perfusion imaging). Without repositioning, the patient was stressed using dipyridamole (0.14mg/kg/min for 5 minutes) with 11 minutes of list mode data acquired starting immediately before the injection of 1122 +/- 170 MBq of tetrofosmin. Both rest and stress injections were delivered mechanically over 30 seconds. A standard set of stress perfusion images were acquired at 45 mins after tracer injection
Arm/Group | Comparision of Myocardial Blood Flow Between PET to SPECT Myocardial Perfusion Imaging.
Number analyzed (Participants) | 31
mean residual difference in MBF | 0.06 (0.37)

2. Primary Outcome: Precision of Myocardial Blood Flow Measurements Between Two SPECT Scans
Description: SPECT myocardial blood flow (MBF) was measured and repeated at a mean interval of 18 days to assess precision of MBF measurements between the two scans.
Time Frame: From enrollment to completion of imaging was a maximum of four weeks.
Population: Patients scheduled for clinically indicated SPECT myocardial perfusion studies who had an intermediate to high pretest probability of disease were 18 years of age or older and had a BMI < 40kg/m2 were recruited to the study.
Measure: Mean (Standard Deviation); unit: % difference in MBF between SPECT scans
Groups:
- Comparison of Myocardial Blood Flow Measurements Between Two SPECT Scans.: Each patient was imaged on two separate occasions using a 1-day rest/stress SPECT MBF protocol. 99mTc-tetrofosmin (370 MBq (2.8 mSv) for rest and 1100 MBq (7.7 mSv) for stress) was delivered using a power injector as a 9 ml bolus over 30 s followed by a 9 ml saline flush over 30 s. Image data was acquired in listmode for 11 min starting just prior to tracer injection. Resting images were acquired first and repeated just prior to stress. For stress, dipyridamole (0.14 mg/kg/min over 5 min) will be given intravenously. At 8 minutes following onset of dipyridamole infusion, stress imaging started prior to the 99mTc-tetrofosmin injection. Aminophylline was administered intravenously at 11 minutes following onset of dipyridamole infusion. The usual post-stress images were acquired approximately 45 minutes after radiotracer injection.
Arm/Group | Comparison of Myocardial Blood Flow Measurements Between Two SPECT Scans.
Number analyzed (Participants) | 30
% difference in MBF between SPECT scans | 29.5 (1.5)

ADVERSE EVENTS:
Time Frame: From enrollment to completion of patient imaging was four weeks.
Description: There was no frequency threshold for reporting adverse events.
Groups:
- Difference Between Measurements of Myocardial Blood Flow Measured With PET and With SPECT: PET studies were acquired with either 82Rb or 13N-ammonia according to clinical protocol. The activity injected at both rest and stress was 10 MBq/kg (82Rb) or 5MBq/kg (ammonia). MBF was based on data acquired over 8 min (82Rb) or 4 min (ammonia). SPECT rest images were obtained for 11 min starting immediately before injection of 316 +/- 71 MBq of 99mTc-tetrofosmin. The patient returned at 45 min after injection for a 5 min static resting acquisition (corresponding to the standard time for myocardial perfusion imaging). Without repositioning, the patient was stressed using dipyridamole (0.14mg/kg/min for 5 minutes) with 11 minutes of list mode data acquired starting immediately before the injection of 1122 +/- 170 MBq of tetrofosmin. Both rest and stress injections were delivered mechanically over 30 seconds. A standard set of stress perfusion images were acquired at 45 mins after tracer injection
Arm/Group | Difference Between Measurements of Myocardial Blood Flow Measured With PET and With SPECT
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT02280941/Prot_SAP_000.pdf